CLINICAL TRIAL: NCT00494689
Title: Transcranial and Rapid Magnetic Stimulation for Gait Apraxia Due to Normal Pressure Hydrocephalus and Cerebral Ischemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Devathasan Neurology Practice Pte Ltd (Other)
Other Study IDs: 02
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2007-07-02 (Estimated); Status verified 2007-06

CONDITIONS: Walking; Cognitive Function
Keywords: transcranial sonolysis or monitoring; rapid magnetic stimulation; cerebral ischemia; hydrocephalus; Barthel's index
MeSH Terms: conditions — Brain Ischemia; Hydrocephalus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigator(neurologist) has published a study in International Congress Series, in the 15th International Conference of Biomagnetism Vancouver Proceedings 2006,and Science Direct website, of 15 patients with brain ischemia and dilated ventricles who improve when treated with transcranial monitoring or low ultrasound wave intensity (milliwatts) and with rapid magnetic stimulation which is also a diagnostic tool routinely used by many neurophysiologists. Before, these patients will progress and may need a brain shunt called Ventriculo-peritoneal shunt. He and collaborators now would like to do a double study as this appears to be a cheap and effective alternative treatment and help patients to walk again.

DETAILED DESCRIPTION:
The transcranial monitoring intensity would be equivalent to the well known CLOTBUST study (<300mw/sq cm)for one hour, using two probes.

All will be treated as an outpatient and there is no form of infusion or interventional treatment.

The rapid magnetic stimulation is at about 50a/us, 15Hz, 1000 pulses with 10 sec pause for ten days along the skull vault. Informed consent will be obtained. 30 patients will be recruited and sham treatment would be just applying probe without power for transcranial and for magnetic stimulation coil will be angled away. Data will be compiled by a separate blinded investigator and so with the statistics. VP shunt failure patients, which is common, will be included. Barthel's daily living index and standard cognitive tests will be used to assess results.

ELIGIBILITY:
Inclusion Criteria:

* cerebral ischemia with our without hydrocephalus and gait apraxia

Exclusion Criteria:

* all other conditions which contribute to walking difficulty e.g. bad knees; or spondylosis; parkinson's or paralytic strokes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-01; Study Completion 2007-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Weng Kiong Aw Yong, Bsc (QUT), Study Chair — Freelancer Computer Programmer and data control
Locations (2):
- Singapore (2):
  - Devathasan Neurology Practice #11-16 MEMC, Singapore
  - Devathasan Neurology Practice, Singapore

REFERENCES:
- [Background] Devathasan G, Dinesh D. Rapid magnetic stimulation with sonolysis for gait apraxia due to to normal pressure hyprocephalus and cerebral ischemia. International Congress Series xx (2007)xxx-xxx( in press)